CLINICAL TRIAL: NCT07355387
Title: Home Based Functional Balance Intervention (FBI) for Physical and Cognitive Symptoms of Multiple Sclerosis
Brief Title: Home Based Functional Balance Intervention for Multiple Sclerosis
Acronym: HomeFBIinMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-0796
Record Dates: First submitted 2025-12-01; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis (MS) - Relapsing-remitting; Multiple Sclerosis (MS) Primary Progressive; Multiple Sclerosis (MS) Secondary Progressive; Multiple Sclerosis Acute and Progressive
Keywords: Home based rehabilitation; Telerehabilitation; Multiple Sclerosis; Mild cognitive impairment; functional balance; safety monitoring; Cognitive motor training; vestibular training
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants assigned to the Functional Balance Intervention (FBI) will complete a 4 month, home based, multicomponent balance and cognitive motor training program. Sessions occur 2 days per week for 1 hour each and are performed independently at home with a designated helper buddy present for safety. Each session includes randomized blocks of functional agility, functional strength, dual task cognitive motor exercises, and vestibular training. Exercises emphasize dynamic balance, multi joint strength, postural control, attention, processing speed, and visuospatial orientation. Dual task components include custom computer based stepping games that integrate cognitive tasks with functional movements. Vestibular components include gaze stabilization, head turn walking, and figure of eight walking. Exercise difficulty progresses based on predefined home evaluation criteria. Participants receive a training manual, home equipment kit, weekly follow up via Zoom, and safety monitoring.
  Interventions: Behavioral: Multicomponent balance intervention consisting of four components including dual-tasking, functional strength, vestibular and dynamic balance.
- Stretching Group (Active Comparator): Participants assigned to the stretching program will complete a 4 month, home based flexibility training regimen matched in duration and frequency to the intervention group. Sessions occur 2 days per week for 1 hour each and include progressive stretching of major upper limb, lower limb, core, and back muscle groups. All stretches are performed in standing to match upright time and positional demands of the Functional Balance Intervention. Each session begins with a brief warm up and concludes with a 10 minute cool down emphasizing relaxation and breathing exercises. Participants receive a printed exercise manual detailing weekly schedules, safety precautions, and instructions for each stretch. No specialized equipment or computer based components are required. A helper buddy must remain present during all sessions for safety. Participants also participate in weekly Zoom check ins to monitor adherence, address concerns, and review home safety recommendations.
  Interventions: Behavioral: Stretching

INTERVENTIONS:
Behavioral: Multicomponent balance intervention consisting of four components including dual-tasking, functional strength, vestibular and dynamic balance. — The Functional Balance Intervention (FBI) is a multicomponent, home based cognitive motor training program designed specifically for persons with Multiple Sclerosis. It integrates four structured constructs-functional agility, functional strength, dual task cognitive motor exercises, and vestibular training-within each 1 hour session. The program uses custom designed interactive dual task stepping games that require simultaneous motor stepping responses and cognitive tasks such as arithmetic, category fluency, and visuospatial cue discrimination. Vestibular components include gaze stabilization, head turn walking, and figure of eight patterns. Progression is individualized using predefined home evaluation criteria (step count, chair stands, tandem stance, single leg stance, and perceived stability). Training is completed independently at home with a helper buddy present and supported by weekly Zoom sessions.
  Arms: Intervention Group
Behavioral: Stretching — The stretching program is a non-progressive, home based flexibility protocol designed to serve as an active control condition. Unlike the Functional Balance Intervention, this program does not include agility, strength, dual task, vestibular, or cognitive motor components, and it does not use computerized games or progressive home evaluations. Participants complete 1 hour sessions, 2 days per week for 4 months, consisting solely of static stretches targeting major upper extremity, lower extremity, trunk, and back muscle groups. All stretches are performed in standing to match the positional demands and session duration of the experimental arm without engaging balance or cognitive systems. The program emphasizes gentle range of motion, posture, breathing, and relaxation rather than neuromotor challenge. No equipment is required beyond the printed stretching manual, and exercises do not progress in complexity or intensity.
  Arms: Stretching Group

SUMMARY:
The study involves a two-arm, Phase 1, randomized controlled clinical trial designed to establish the feasibility and effects of a Functional Balance Intervention (FBI) on physical and cognitive function, as well as measures of daily living among persons with multiple sclerosis (PwMS).

Combined Specific Aims:

Aim 1: Examine the effect of the FBI (Intervention Group) on physical function in PwMS compared to a stretching program (Control Group).

Hypothesis 1: After four months of training, the FBI group will show significantly greater improvements in physical function compared to the stretching group.

Aim 2: Examine the effect of the multicomponent FBI on cognitive function in PwMS compared to the stretching program.

Hypothesis 2: After four months of training, the FBI group will show significantly greater improvements in cognitive function compared to the stretching group.

Aim 3: Examine the effects of the multicomponent FBI compared to the Control Group among PwMS on measures of daily living (dual-task performance, balance confidence, community mobility, and quality of life).

Hypothesis 3: After four months of training, the FBI group will show significantly greater improvements in measures of daily living compared to the stretching group.

All assessment sessions will be conducted virtually via Zoom. All measures collected during the initial screening, pre-training assessment, training progression, and mid- and post-training assessment sessions will be administered either via Zoom with a Helper Buddy present or through survey links sent to participants via the UIC REDCap system. The training sessions will be performed independently by the participants in the presence of a Helper Buddy.

The investigators will recruit 75 people with multiple sclerosis (PwMS) for this study. Eligible participants will be randomized to either the FBI (Intervention) or stretching (Control) group, followed by an onboarding session with a designated Helper Buddy. Training will occur twice weekly for four months. Based on the anticipated attrition rate, the investigators aim for 40 PwMS to complete the post-training assessments and finish the study.

DETAILED DESCRIPTION:
This project investigates the feasibility of a remote, home-based Functional Balance Intervention (FBI) targeting the physical and cognitive symptoms of multiple sclerosis (MS).

The study is a two-arm, Phase 1, randomized controlled clinical trial designed to establish the feasibility and effects of the FBI on physical and cognitive function, as well as measures of daily living among persons with multiple sclerosis (PwMS). Because the exercise training will be completed independently at home, additional precautionary measures for participant safety (such as requiring a Helper Buddy) and modified home evaluations will be implemented to monitor training progression.

A total of 75 people with multiple sclerosis (PwMS) will be recruited and undergo a telephone screening. Accounting for an estimated 20% screening failure rate, the investigators expect to enroll approximately 60 PwMS in the project. Based on an additional 20% expected attrition following the initial screening, approximately 48 PwMS are anticipated to be eligible for participation. Eligible participants will complete one pre-training assessment session before being randomized into one of two groups: the FBI (Intervention Group) or the Stretching (Control) group.

Following randomization, each participant and their designated Helper Buddy will complete an onboarding session that provides detailed instructions regarding assessment procedures and training logistics. Participants will then engage in independent training sessions with their Helper Buddy twice per week for four months. Given the expected 15-17% attrition rate based on prior experience, the target final sample size is 40 PwMS. The investigators expect 40 participants to complete post-training assessments after four months and finish the study.

All assessment sessions will be conducted virtually via Zoom. Measures collected during the initial screening, pre-training assessment, training progression checks, and post-training assessment will occur either via Zoom with a Helper Buddy present or through survey links distributed via the University of Illinois REDCap system. Training sessions will be performed independently by participants in the presence of their Helper Buddy.

The overall goal of this project is to determine the feasibility of the FBI and evaluate its impact on physical and cognitive functions, as well as other measures of daily living among PwMS in a home-based environment. This protocol builds on strong evidence from previous successful trials involving neurological populations. It has been piloted in a laboratory setting with individuals with stroke and mild cognitive impairment, demonstrating both safety and efficacy. In addition, it has been tested in telerehabilitation formats among healthy older adults and frail older individuals, with results indicating feasibility, safety, and effectiveness for independent home exercise and no reported adverse events.

The investigators now intend to translate this evidence-based protocol to examine its effects in people with multiple sclerosis. If successful, this study could have substantial impact by providing a low-cost, safe, and effective intervention that increases accessibility for rural and underserved populations.

ELIGIBILITY:
Inclusion Criteria

Telephone Screening Inclusion Criteria:

1. Age 40-90 years.
2. Self-reported diagnosis of Multiple Sclerosis.
3. On stable disease-modifying therapy for ≥6 months.
4. No PT/OT balance-related therapy in the past 6 months.
5. Able to stand from a chair independently (with or without hand support).
6. Score 25-75% on the 12-item MS Walking Scale.
7. No other neurological, cardiopulmonary, musculoskeletal, or systemic conditions affecting standing/walking.
8. English speaking.
9. Willing to complete all study procedures including Zoom sessions.
10. Has reliable internet access.
11. Has a helper buddy available for all sessions.
12. Possible mild cognitive impairment based on self-report.

Initial Screening Inclusion Criteria:

1. Moderate disability: ePR-EDSS score 4.0-6.5.
2. Mild cognitive impairment: MoCA 18-25, or Jak/Bondi criteria for those scoring 26-30.
3. Physically inactive or moderately active (Godin score <24).
4. Cardiovascular safety parameters within acceptable limits.
5. No global aphasia (Mississippi Aphasia Screening Test ≥71 percent).
6. Berg Balance Scale score ≥40/56.
7. Able to walk 1 block with or without an assistive device.

Helper Buddy Inclusion Criteria:

1. Age ≥18 years.
2. Lives within close proximity to the participant.
3. No self-reported major medical conditions limiting safety assistance.
4. English speaking.
5. Able to attend all training and assessment sessions.
6. Able to assist with basic safety, positioning, and communication with the research team.
7. Has internet access and can use Zoom.

Exclusion Criteria

Telephone Screening Exclusion Criteria:

1. MS relapse or exacerbation within the past 3 months.
2. Recent major surgery (<6 months) or hospitalization (<3 months).
3. Resting shortness of breath or uncontrolled pain >3/10.
4. Uncontrolled hypertension or diabetes.
5. Bone fracture in the past 6 months.
6. Disability limiting activities of daily living.
7. History of epilepsy or uncontrolled seizures in past year.
8. Sedative medication use that may interfere with training.
9. Use of Alzheimer's/dementia-modifying drugs or enrollment in AD clinical trials.
10. Use of antidepressants or anxiety medications.
11. Moderate or high risk on PAR-Q (≤1 "yes" response).
12. Severe cognitive impairment (TICS-M ≥18).
13. Currently receiving cognitive or physical rehabilitation.
14. Pacemaker use.

Initial Screening Exclusion Criteria:

1. Cardiovascular parameters outside safety limits (HR, BP, O₂ saturation).
2. Global aphasia (Mississippi <71 percent).
3. Peripheral nerve injury.
4. Berg Balance Scale <40/56.
5. Inability to walk one block with or without an assistive device.

Population Exclusions:

1. Non-English speakers (protocol delivered only in English).
2. Individuals under 18 years.
3. Pregnant individuals.
4. Prisoners or other vulnerable populations.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-11-24 (Estimated); Study Completion 2027-11-24 (Estimated)

PRIMARY OUTCOMES:
Safety: occurrence of adverse events | Last week of training (Month 4)
  Non-serious adverse events may include transient muscle soreness, fatigue, mild dizziness, temporary loss of balance corrected by the helper buddy, or minor joint discomfort during home exercise. These events do not require medical intervention and are reported during weekly check ins or directly to study staff.
  Serious adverse events include any event resulting in injury requiring medical care, hospitalization, life-threatening symptoms, severe cardiovascular responses (chest pain, uncontrolled shortness of breath, hypertensive crisis), oxygen desaturation below safety thresholds, or falls causing significant injury. The helper buddy is instructed to stop activity immediately, call emergency services when necessary, and notify the research team.
  All adverse events are monitored throughout screening, assessments, and training sessions, and are reviewed by the PI with prompt IRB reporting as required.
Adherence | End of training (Month 4)
  Adherence will be monitored by tracking completion of all scheduled home training sessions, weekly Zoom check ins, and timely completion of progression evaluations and questionnaires. Participants are expected to complete 2 sessions per week for 4 months, and adherence will be defined as completing at least 75 percent of planned sessions. Attendance logs, helper buddy confirmation, and participant self reports are reviewed weekly by study staff to document adherence and address barriers to participation.
Change in Physical Function measured by Short Physical Performance Battery | Baseline, 1 week post-training
  The Short Physical Performance Battery (SPPB) is a validated measure of lower extremity physical function that includes three components: standing balance, gait speed, and repeated chair stands. Balance is assessed using side by side, semi tandem, and tandem stances; gait speed is measured over a short walking distance; and strength/mobility is evaluated using five repeated chair rises. Scores from each component are combined into a 0-12 total score, with higher scores indicating better physical function. For this study, the SPPB is administered remotely over Zoom with camera positioning and helper buddy support to ensure safety during all standing and mobility tasks.
Change in Walking Function: Dynamic Gait Index (DGI) | Baseline, 1 week post-training
  The Dynamic Gait Index (DGI) is a clinical measure of functional gait performance that assesses an individual's ability to adapt walking to varying task demands. The test includes eight walking tasks such as changing gait speed, head turns, pivot turns, stepping over obstacles, and stair climbing. Each task is scored on a 0-3 scale, with a maximum total score of 24; higher scores indicate better dynamic gait stability. In this study, the DGI is administered remotely with helper buddy supervision to ensure safety during all gait tasks.
Change in Walking endurance: Timed 25-Foot Walk | Baseline, 1 week post-training
  The Timed 25-Foot Walk is a standardized measure of gait speed and lower extremity mobility in persons with neurological conditions. Participants are instructed to walk 25 feet as quickly and safely as possible, and the time to complete the distance is recorded in seconds. Faster times indicate better ambulatory function. In this study, the Timed-25 Foot Walk is administered remotely over Zoom with appropriate camera positioning and helper buddy supervision to ensure safety during the walking task.
Change in information processing speed | Baseline, 1 week post-training
  The Symbol Digit Modalities Test evaluates information processing speed, attention, and visual scanning. Participants are shown a key that pairs simple symbols with numbers and are asked to verbally report the number corresponding to each symbol presented on the screen as quickly and accurately as possible within a fixed time period. The test takes approximately 5 minutes to complete. The Symbol Digits Modalities score is calculated as the total number of correct symbol-number pairings completed within the time limit, with scores typically ranging from 0 to approximately 110. Higher scores indicate faster processing speed and better performance, while lower scores reflect greater difficulty with information processing.
Change in verbal learning and memory | Baseline, 1 week post-training
  The California Verbal Learning Test-II assesses verbal learning and memory. Participants hear a list of words read aloud by the examiner and are asked to recall as many words as possible immediately after each presentation. This procedure is repeated across five learning trials using the same word list. The task takes approximately 7-10 minutes. The score used for BICAMS is the total number of words correctly recalled across the five learning trials, with possible scores ranging from 0 to 80. Higher scores indicate better verbal learning and memory, while lower scores indicate greater difficulty with learning and recalling verbal information.
Change in visuospatial learning and memory | Baseline, 1 week post-training
  The Brief Visuospatial Memory Test-Revised evaluates visuospatial learning and memory. Participants are briefly shown a display of simple geometric figures arranged in a specific pattern. After the figures are removed, participants are asked to reproduce the figures and their locations from memory. This process is repeated across three learning trials and takes approximately 5 minutes. The Brief Visuospatial Memory Test-Revised score used for Brief International Cognitive Assessment for Multiple Sclerosis is the total recall score across the three trials, with possible scores ranging from 0 to 36. Higher scores indicate better visuospatial learning and memory, while lower scores reflect greater visuospatial memory impairment.
Change in Dual-task balance cost | Baseline, 1 week post-training
  Dual-Task Balance Cost (Limits of Stability + Letter-Number Sequencing) Dual-task balance cost is assessed by combining the Limits of Stability test with a concurrent Letter-Number Sequencing task. Participants perform controlled reaching movements in multiple directions while simultaneously generating an alternating number-letter sequence. Balance performance (reach distance and control) and cognitive accuracy are recorded under both single-task and dual-task conditions. Dual-task cost is calculated as the relative change in balance performance when the cognitive task is added. This assessment is conducted remotely over Zoom with helper buddy supervision for safety.
Change in Community Mobility: University of Alabama Birmingham (UAB) Questionnaire | Baseline, 1 week post-training
  The Life-Space Questionnaire assesses real-world community mobility by capturing how far and how often a person moves through different life-space levels, ranging from within the home to travel outside the local community. Scores reflect the frequency, independence, and distance of mobility over the past four weeks, with higher scores indicating greater community mobility. In this study, the questionnaire is completed remotely via REDCap or Zoom based on participant preference.
Change in Community Mobility: Accelerometer | Baseline, 1 week post-training
  Community mobility is objectively measured using a wearable ActiGraph accelerometer worn for 7 consecutive days for at least 12 hours per day. The device captures step counts, activity levels, and movement patterns that reflect real-world mobility outside the laboratory or home. Data are downloaded and analyzed to quantify overall mobility and time spent in different activity intensities. Participants receive the device by mail and return it using a prepaid shipping label.
Change in Quality of Life: Multiple Sclerosis Impact Scale (MSIS-29) | Baseline, 1 week post-training
  Quality of life is assessed using the Multiple Sclerosis Impact Scale (MSIS-29), a validated self-report questionnaire measuring the physical (20 items) and psychological (9 items) impact of MS on daily functioning. Scores reflect the extent to which MS affects mobility, activities, mood, and overall well-being, with higher scores indicating greater impact. The MSIS-29 is completed remotely via REDCap or during a Zoom session based on participant preference.
Change in Balance Confidence: Activities-Specific Balance Confidence (ABC) | Baseline, 1 week post-training
  Balance confidence is measured using the Activities-Specific Balance Confidence (ABC) Scale, a validated 16-item questionnaire assessing an individual's confidence in performing common daily activities without losing balance. Participants rate their confidence from 0 to 100 percent for each activity, with higher scores indicating greater balance self-efficacy. The ABC Scale is completed remotely via REDCap or during a Zoom session according to participant preference.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains identifiable health information collected through remote assessments, cognitive testing, and video-based evaluations. Given the nature of home-based balance and mobility data, full de-identification cannot be guaranteed, and the IRB does not permit external sharing of raw video or sensor-based data. Summary results will be shared in publications and presentations, but IPD will not be made available.

REFERENCES:
- [Background] Kannan L, Vora J, Bhatt T, Hughes SL. Cognitive-motor exergaming for reducing fall risk in people with chronic stroke: A randomized controlled trial. NeuroRehabilitation. 2019;44(4):493-510. doi: 10.3233/NRE-182683. PMID 31256084
- [Background] Tramontano M, Martino Cinnera A, Manzari L, Tozzi FF, Caltagirone C, Morone G, Pompa A, Grasso MG. Vestibular rehabilitation has positive effects on balance, fatigue and activities of daily living in highly disabled multiple sclerosis people: A preliminary randomized controlled trial. Restor Neurol Neurosci. 2018;36(6):709-718. doi: 10.3233/RNN-180850. PMID 30412513
- [Background] Veldkamp R, Baert I, Kalron A, Tacchino A, D'hooge M, Vanzeir E, Van Geel F, Raats J, Goetschalckx M, Brichetto G, Shalmoni N, Hellinckx P, De Weerdt N, De Wilde D, Feys P. Structured Cognitive-Motor Dual Task Training Compared to Single Mobility Training in Persons with Multiple Sclerosis, a Multicenter RCT. J Clin Med. 2019 Dec 10;8(12):2177. doi: 10.3390/jcm8122177. PMID 31835502
- [Background] DeLuca J, Chiaravalloti ND, Sandroff BM. Treatment and management of cognitive dysfunction in patients with multiple sclerosis. Nat Rev Neurol. 2020 Jun;16(6):319-332. doi: 10.1038/s41582-020-0355-1. Epub 2020 May 5. PMID 32372033
- [Background] Motl RW, Sandroff BM, Kwakkel G, Dalgas U, Feinstein A, Heesen C, Feys P, Thompson AJ. Exercise in patients with multiple sclerosis. Lancet Neurol. 2017 Oct;16(10):848-856. doi: 10.1016/S1474-4422(17)30281-8. Epub 2017 Sep 12. PMID 28920890